CLINICAL TRIAL: NCT05880043
Title: An Open-label, Multi-center, Dose-escalation and Expansion, Phase 1/2a Study to Evaluate the Safety, Tolerability, PK/PD, and Preliminary Anti-tumor Activity of GIC-102 Monotherapy in Patients With Advanced Solid Tumors, R/R Non-Hodgkin Lymphoma, and Multiple Myeloma
Brief Title: GIC-102, Intravenous Allogeneic NK Cells, in Subjects With Advanced Solid Cancers and R/R Hematologic Malignancies
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: GI Cell, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GIC-102101
Record Dates: First submitted 2023-04-24; First posted 2023-05-30 (Actual); Last update posted 2024-07-09 (Actual); Status verified 2024-06

CONDITIONS: Advanced Solid Tumors; Relapsed/Refractory Non-Hodgkin Lymphoma; Relapsed/Refractory Multiple Myeloma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Multiple Myeloma

STUDY DESIGN:
Intervention Model Description: Dose escalation phase: up to 30 subjects / Dose expansion phase: up to 20 subjects
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dose escalation phase: GIC-102 monotherapy (Experimental): * Low Dose level 1: 1 x 10^9 cells
  * Mid Dose level 2: 3 x 10^9 cells
  * High Dose level 3: 1 x 10^10 cells
  Interventions: Drug: GIC-102
- Dose expansion phase: GIC-102 monotherapy (Experimental): - Dose level: RP2D
  Interventions: Drug: GIC-102

INTERVENTIONS:
Drug: GIC-102 — GIC-102 will be administered via IV infusion 3 times at intervals of 1 week, and 28 days is defined as 1 cycle
  Arms: Dose escalation phase: GIC-102 monotherapy
Drug: GIC-102 — GIC-102 will be administered via IV infusion 3 times at intervals of 1 week, and 28 days is defined as 1 cycle
  Arms: Dose expansion phase: GIC-102 monotherapy

SUMMARY:
This is a first-in-human trial to investigate the safety, tolerability, pharmacokinetics, pharmacodynamics, and antitumor effects of GIC-102 in patients with advanced solid tumors, relapsed/refractory non-hodgkin lymphoma, and multiple myeloma.

DETAILED DESCRIPTION:
This is a first-in-human, open-label, non-randomized, dose-escalation and expansion phase 1/2a trial to determine the safety profile and identify the maximum tolerated dose of GIC-102 in patients with advanced solid tumors, relapsed/refractory non-hodgkin lymphoma, and multiple myeloma.

This study will comprise two phases.

* GIC-102 monotherapy dose escalation Phase
* GIC-102 monotherapy dose expansion phase

GIC-102 is an "off-the-shelf" allogeneic natural killer cells isolated from non-HLA-related healthy donor. Natural killer cells are innate immune cells that show strong cytolytic function against physiologically stressed cells such as tumor cells and virus infected cells.

ELIGIBILITY:
Inclusion criteria:

1. At least 19 years of age
2. Advanced solid tumors, relapsed/refractory non-hodgkin lymphoma, and multiple myeloma
3. At least one measurable or evaluable lesion
4. Eastern Cooperative Oncology Group performance status 0 or 1
5. A life expectancy of 12 weeks or more
6. Acceptable hematological function, kidney, and liver function
7. Subjects who sign on an informed consent form willingly

Exclusion Criteria:

1. Clinically significant cardiovascular disease within 24 weeks
2. Primary malignant tumor other than the indications for this study
3. The following diseases

   1. Severe infection or other uncontrolled active infectious disease requiring administration of systemic antibiotics or antivirals within 4 weeks
   2. The New York Heart Association class III/IV
   3. Active hepatitis B virus or hepatitis C virus infection
   4. Human immunodeficiency virus positive
   5. Clinically significant symptoms or uncontrolled central nervous system metastasis
4. Previously been diagnosed with immunodeficiency or need systemic corticosteroids or other systemic immunosuppressants within 2 weeks or require administration of systemic immunosuppressants during the study
5. Received chemotherapy other than pre-conditioning within 4 weeks
6. Underwent major surgery within 4 weeks prior or minor surgery within 2 weeks
7. Hypersensitivity reactions to the study drug or excipients
8. Hypersensitivity to cyclophosphamide or fludarabine
9. Have received allogeneic cell therapy within 6 months or autologous stem cell therapy within 4 weeks
10. Have previously received an allogeneic tissue/solid organ transplant
11. Have administered other investigational drug or applied other investigational medical device within 4 weeks
12. Pregnant or lactating female subjects
13. Male subjects who did not agree to use contraception or to maintain abstinence

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-04-28 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicity assessment (dose escalation phase) | Up to 4 weeks
  To determine the maximum tolerated dose of allogeneic natural killer cells
Adverse event / Immune related adverse event | through study completion, an average of 1 year
  To determine the safety of GIC-102
Objective Response Rate (ORR) (dose expansion phase) | through study completion, an average of 1 year
  To evaluate the efficacy of GIC-102 according to RECISTv1.1(solid tumor), Lugano 2014 (non-Hodgkin's lymphoma), IMWG 2016 (multiple myeloma)

SECONDARY OUTCOMES:
Objective response rate (ORR) (dose escalation phase) | through study completion, an average of 1 year
  To evaluate the efficacy of GIC-102 according to RECISTv1.1(solid tumor), Lugano 2014 (non-Hodgkin's lymphoma), IMWG 2016 (multiple myeloma)
Progression free survival (PFS) | Through study completion / 6-month, 12-month, 18-month (solid tumor, dose expansion phase)
  Duration from start of study treatment to progression diease or death (regardless of cause), whichever comes first
Overall survival (OS) | Through study completion / 6-month, 12-month, 18-month, overall timepoint(dose expansion phase)
  Duration from start of study treatment to death (regardless of cause)
Duration of response (DOR) | Through study completion
  Time from the first occurrence of a documented objective response to the time of the first document disease progression or death from any cause
Disease Control Rate (DCR) | through study completion, an average of 1 year
  Percentage of patients who have achieved CR, PR and stable disease (SD)
PK Profile (dose expansion phase) -Cmax | up to 6 months
PK Profile (dose expansion phase) - Tmax | up to 6 months
PK Profile (dose expansion phase) - AUC | up to 6 months

OTHER OUTCOMES:
PK Profile (dose escalation phase) -Cmax | up to 6 months
PK Profile (dose escalation phase) - Tmax | up to 6 months
PK Profile (dose escalation phase) - AUC | up to 6 months
Immune Profile | through study completion, an average of 1 year
  * Immune response activation factor (Immune subset marker, cytokine expression)
  * Immunophenotyping of peripheral blood mononuclear cells will be performed by flow cytometry
Alloantibody Identification | through study completion, an average of 1 year
  * donor human leukocyte antigen (HLA) class I-specific antibody (positive/negative)
  * donor HLA class II-specific antibody (positive/negative)

CONTACTS AND LOCATIONS:
Locations (3):
- South Korea (3):
  - Korea University Anam Hospital, Seoul
  - Seoul Asan Medical center, Seoul
  - Seoul National University Hospital, Seoul

IPD SHARING:
Plan to Share IPD: No